CLINICAL TRIAL: NCT00002315
Title: A Double-Blind, Multicenter Study Comparing Oral 882C87 With Oral Acyclovir for Treatment of Localized Herpes Zoster in Immunocompromised Patients
Brief Title: A Comparison of 882C87 Versus Acyclovir in the Treatment of Herpes Zoster in Patients With Weakened Immune Systems
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 130A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-05

CONDITIONS: HIV Infections; Chickenpox
Keywords: Herpes Zoster; Acyclovir; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Chickenpox; Herpes Zoster; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — 5-propynylarabinofuranosyluracil; Acyclovir

INTERVENTIONS:
Drug: Netivudine
Drug: Acyclovir

SUMMARY:
To determine the efficacy of oral 882C87 compared with oral acyclovir in the treatment of localized herpes zoster in immunocompromised patients. To assess the safety and tolerance of oral 882C87 in immunocompromised patients.

DETAILED DESCRIPTION:
Patients are randomized to receive either 882C87 or acyclovir with corresponding placebos for 14 days, with two hundred patients in each of the two groups. They are stratified by presence or absence of HIV infection. Patients undergo 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Acute localized herpes zoster or rash present less than 72 hours, verified by clinical diagnosis.
* Immunocompromised condition primarily as a result of documented HIV infection, malignancy, chemotherapy or radiation therapy, solid organ or bone marrow transplant, or chronic immunosuppressive therapy.
* Life expectancy of at least 6 months.
* Ability to cooperate with the requirements of the study.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Evidence of cutaneous or visceral dissemination (more than 20 discrete lesions outside adjacent dermatomes).
* Acute, life-threatening condition.
* Significant malabsorption syndrome or other gastrointestinal dysfunction that may severely reduce drug absorption.
* Intolerance of oral medication.

Concurrent Medication:

Excluded:

* Tricyclic antidepressants or anti-epileptics.
* Topical applications to the zoster lesions that would obscure evaluation.
* Fluorouracil and flucytosine.
* Systemic therapy with agents with antiherpetic activity (from 2 weeks prior to first dose to day 28 of study).
* Probenecid or other drugs likely to affect elimination of study drugs (from 2 days prior to first dose to day 14 of the study).
* Capsaicin (Zostrix).
* Warfarin (Coumadin) during 14 days of treatment.

Patients with the following prior conditions are excluded:

History of intolerance, hypersensitivity, or severe drug reaction to acyclovir.

Prior Medication:

Excluded:

* Systemic therapy with agents with antiherpetic activity (including interferon) within the past 2 weeks.
* Probenecid or other drugs likely to affect the elimination of 882C87 or acyclovir within the past 48 hours.
* Drugs likely to interact with 882C87 (e.g., fluorouracil or flucytosine) within the past 7 days.
* Zoster immune globulin or zoster immune plasma within the previous month. History of alcohol or drug abuse within the previous 6 months or current methadone therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Simon - Williamson Clinic, Birmingham, Alabama
  - SORRA / NC Research Ctr, Birmingham, Alabama
  - Univ of Arizona / Univ Med Ctr, Tucson, Arizona
  - Cedars Sinai Med Ctr, Los Angeles, California
  - AIDS Community Research Consortium, Redwood City, California
  - Saint Francis Mem Hosp, San Francisco, California
  - Sunnyvale Med Clinic, Sunnyvale, California
  - Clinical Research Consultants, Trumbull, Connecticut
  - Med Associates Clinic, Dubuque, Iowa
  - Oschner Clinic, New Orleans, Louisiana
  - Washington Univ, St Louis, Missouri
  - New Mexico Med Group, Albuquerque, New Mexico
  - Jordon Diagnostics and Research Inc, High Point, North Carolina
  - Hanover Med Specialists, Wilmington, North Carolina
  - Oregon Research Group, Eugene, Oregon
  - Oregon Health Sciences Univ, Portland, Oregon
  - Roger Williams Med Ctr, Providence, Rhode Island
  - Silver Lake Med Inc, Providence, Rhode Island
  - Vanderbilt Med Ctr, Nashville, Tennessee
  - N Texas Ctr for AIDS & Clin Rsch, Dallas, Texas
  - MacGregor Med Association, Houston, Texas
  - Univ TX Med Branch, Nassau Bay, Texas
  - Infections Ltd / Physicians Med Ctr, Tacoma, Washington
  - Med Consultants LTD, Milwaukee, Wisconsin
  - Rhinelander Med Ctr, Rhinelander, Wisconsin